CLINICAL TRIAL: NCT06846996
Title: Real-world Effectiveness and Safety of Trastuzumab Deruxtecan in Patients With Locally Advanced or Metastatic HER2-positive Gastric or Gastroesophageal Junction Adenocarcinoma in China: A Nation-wide, Multi-center, Prospective, Non-interventional Study
Brief Title: Real-world Effectiveness and Safety of Trastuzumab Deruxtecan in Patients With Locally Advanced or Metastatic HER2-positive Gastric or Gastroesophageal Junction Adenocarcinoma in China
Acronym: RECOVER
Status: Recruiting | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: DS8201-0076-NIS-MA
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: HER2-positive Gastric Cancer; HER2-positive Gastroesophageal Junction
Keywords: HER2-positive gastric cancer; HER2-positive gastroesophageal junction
MeSH Terms: interventions — trastuzumab deruxtecan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HER2-positive gastric/gastroesophageal junction adenocarcinoma: Patients who are diagnosed with locally advanced or metastatic HER2-positive gastric or gastroesophageal junction adenocarcinoma who made a decision (prior to enrolling in this study) to receive T-DXd treatment in a clinical practice setting.
  Interventions: Drug: Trastuzumab deruxtecan (T-DXd)

INTERVENTIONS:
Drug: Trastuzumab deruxtecan (T-DXd) — This is an non-interventional, observational study. No drug will be provided or administered as part of this protocol; however, participants on T-DXd (starting dose 6.4 mg/kg IV Q3W) will be enrolled in this study as part of clinical routine or the clinical judgement of physician.

SUMMARY:
Trastuzumab deruxtecan's (T-DXd's) efficacy and safety has been confirmed in traditional clinical trials, there is a lack of real-world evidence, especially among Chinese patients. The objective of this study is to evaluate real-world effectiveness and safety profile of T-DXd by collecting real-world data treating in patients with locally advanced or metastatic HER2-positive gastric or gastroesophageal junction adenocarcinoma.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the effectiveness of T-DXd in real-world setting (real-word time to treatment failure).

The secondary objectives of this study are to assess the safety profile of T-DXd (treatment related adverse events [TRAE] regardless of grade, and physician reported adverse events of special interest [AESI] regardless of grade, etc.) and to evaluate effectiveness of T-DXd (real-world time to next treatment). This is an non-interventional, observational study. No drug will be provided or administered as part of this protocol; however, participants on T-DXd will be enrolled in this study.

ELIGIBILITY:
Participants must meet all the following inclusion criteria to be eligible for the study:

1. Participants with pathologically diagnosed locally advanced unresectable or metastatic gastric cancer/gastroesophageal junction adenocarcinoma (GC/GEJA).
2. ≥18 years of age at the time of starting the first dose of T-DXd and signing informed consent form (ICF), capable of providing informed consent.
3. HER2-positive status (IHC 3+ or IHC 2+/ISH +).
4. Received prior anti-cancer treatment regimens according to National Medical Products Administration indication or clinical judgement of physician.
5. Decision to newly initiate T-DXd before study ICF signing. If the participants have started the first dose of T-DXd no longer than 21 days before enrollment, they could be enrolled if the signed and dated ICF could be obtained.

Exclusion Criteria：

Participants who meet any of the following criteria will be excluded from the study:

1. Pregnancy or breastfeeding.
2. Participants who at the time of data collection of the study are participating in or have participated in an interventional study that remains blinded.
3. Known hypersensitivity to either the drug substances or inactive ingredients in the drug product.
4. Judged by the investigator to be unfit to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants for this study include participants with HER2-positive local advanced or metastatic GC/GEJA.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Real-world Time to Treatment Failure (rwTTF) | T-DXd treatment initiation date (index date) to date of treatment discontinuation due to disease progression, physician decision, adverse events or death, whichever occurs first, up to approximately 2 years
  rwTTF is defined as time from T-DXd treatment initiation date to the earliest date of treatment discontinuation due to disease progression, physician decision, adverse events or death.

SECONDARY OUTCOMES:
Number of Participants Reporting Treatment Related Adverse Events (TRAE) and Physician-reported Adverse Event of Special Interest (AESI), Regardless of Grade | T-DXd treatment initiation date (index date) until end of study, or death, or withdrawal of consent, or loss to follow-up (LTFU), or study closure, whichever occurs first, up to approximately 2 years
  A TRAE is defined as a harmful reaction, resulting from the normal usage and dosage to a medicinal product, which is unrelated to the purpose of medication. Physician-reported AESIs are defined as interstitial lung disease/pneumonitis and left ventricular ejection fraction decrease.
Real-world Time to Next Treatment (rwTTNT) | T-DXd treatment initiation date (index date) to the date of receiving next line anti-cancer treatment or death, whichever occurs first, up to approximately 2 years
  rwTTNT is defined as time from T-DXd treatment initiation date to the earliest date of receiving next line anti-cancer treatment, or death.

CONTACTS AND LOCATIONS:
Overall Officials: Project Manager, Study Director — Daiichi Sankyo Co., Ltd.
Locations (36):
- China (36):
  - China-Japan Friendship Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - Beijing GoBroad Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Changzhi People's Hospital, Changzhi
  - Fujian Cancer Hospital, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou
  - Guangdong Hospital of Traditional Chinese Medicine, Guangzhou
  - Hainan General Hospital, Haikou
  - Zhejiang Cancer Hospital, Hangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Anhui Province Cancer Hoospital, Hefei
  - Jiangmen Central Hospital, Jiangmen
  - Nanjing Drum Tower Hospital, Nanjing
  - Jiangsu Cancer Hospital, Nanjing
  - Shanghai GoBroad Cancer Hospital, Shanghai
  - Shanghai ninth People's Hospital,Shanghai Jiaotong University School of Medicine, Shanghai
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Zhongshan Hospital, Shanghai
  - Huadong Hospital Affiliated to Fudan University, Shanghai
  - Cancer Hospital of Shantou University Medical College, Shantou
  - Liaoning Cancer Hospital, Shenyang
  - Shanxi Cancer Hospital, Taiyuan
  - Taizhou Hospital of Zhejiang Province, Taizhou
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - The Second Hospital of Tianjin Medical University, Tianjin
  - The Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Affiliated Hospital of Xiamen University, Xiamen
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No